CLINICAL TRIAL: NCT01168167
Title: Comparing the Dynamics of Different HIV-1 cDNA Species in CD4-positive T-cells and HIV-1 RNA in Plasma of Infected Individuals After Initiation of Antiretroviral Therapy With or Without Raltegravir
Brief Title: Impact of Raltegravir on HIV-1 cDNA Slope Following Antiretroviral Therapy (ART) Initiation
Status: Completed | Type: Observational
Sponsor: Christoph Stephan (Other)
Collaborators: University Hospital Heidelberg (Other)
Responsible Party: Sponsor-Investigator, Christoph Stephan, Professor, Goethe University
Organization: Goethe University (Other)
Other Study IDs: JWG-HIVCENTER-Hopp1
Record Dates: First submitted 2010-07-21; First posted 2010-07-23 (Estimated); Last update posted 2016-03-23 (Estimated); Status verified 2016-03

CONDITIONS: HIV-1
Keywords: Antiretroviral Therapy, Highly Active; MK 0518; HIV-1 DNA species; viral slope; Ribonucleic Acid; DNA, Complementary

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- raltegravir-based cART: Patients who begin cART in regular clinical routine with 2N(t)RTI plus raltegravir (n=10 patients) will be offered to participate in this observation arm, but only if no other antiretroviral drugs and no concomitant drugs with relevant impact on antiretroviral's pharmacokinetics are administered. At time of study inclusion, patients should be characterised by a HIV-1 RNA load of >5,000 copies/mL and CD4-cell count of >200/µL within 12 weeks before cART initiation.
- standard of care-cART: Patients who begin cART in regular clinical routine with 2N(t)RTI plus either a boosted protease inhibitor or efavirenz (n=10 patients) at standard doses will be offered to participate in this observation arm. They will be offered to participate in this trial only if no other antiretroviral drugs and no concomitant drugs with relevant impact on antiretroviral's pharmacokinetics are administered. At time of study inclusion, patients should be characterised by a HIV-1 RNA load of >5,000 copies/mL and CD4-cell count of >200/µL within 12 weeks before cART initiation.

SUMMARY:
Recent clinical trials of combination antiretroviral therapy (cART) containing the first approved integrase inhibitor (i.e. raltegravir) have demonstrated a more rapid decay of HIV-1 RNA in plasma, compared to conventional potent antiretroviral combinations. This was observed especially during the early phase (up to week 12) following initiation of cART.

To explain this, two mechanistic hypotheses have been developed:

1. - Macrophage reservoir death hypothesis. A major source of virus production during the second phase decay are believed to be long-lived infected cells with continuous virus production - e.g. macrophages. An accumulation of unintegrated, episomal HIV-1 cDNAs can promote apoptosis (Li et al. Embo J. 2001;20: 3272). In case of HIV superinfection of such a productively infected cell, an INI-based cART may induce apoptosis and thus contribute to a decrease in HIV RNA load during second phase decay. However, no study has thus far addressed the consequences of INI treatment on HIV-1 cDNA species on any cell population in vivo.
2. - Resting CD4 T-cell reservoir integration block hypothesis. Resting CD4 T-cells may represent a substantial reservoir for HIV replication during the second phase decay as well. A special characteristic of these cells is that HIV-1 cDNA is typically localized to the nucleus in a not-integrated form (Chun et al., PNAS 1997;94:13193). These resting cells likely integrate HIV-DNA upon activation and then contribute to HIV viremia and viral spread. Conceptually, integration could be prevented by RGV, but not by RTI or PI. An accumulation of circular episomal HIV-1 cDNA species may also be a consequence of RGV treatment in this cell type.

Patient disposition:

To explore raltegravir-induced shifts in HIV-1 cDNA species in vivo, this non-interventional clinical observation investigates the dynamics of the three major HIV-1 cDNA species (total HIV-1 cDNA, HIV-1 integrants in the host cell genome, episomal HIV-1 2-LTR circles) over a period of 4 months in two groups of patients starting off cART from a single study center. Patients who begin cART in regular clinical routine with 2N(t)RTI plus either (n=10 patients) raltegravir or (n=10 patients) a boosted protease inhibitor/ alternatively an NNRTI will be offered to participate in this observation. Only patients are offered to participate in this trial if no other antiretroviral drugs than the above mentioned and no concomitant drugs with relevant impact on antiretroviral's pharmacokinetics are administered. At time of study inclusion, patients should be characterised by a HIV-1 RNA load of >5,000 copies/mL and CD4-cell count of >200/µL within 12 weeks before cART initiation.

Preliminary analyses of PBMCs from HIV-infected patients indicate that all three major HIV-1 cDNA species can be quantified by real-time PCR under these baseline conditions.

ELIGIBILITY:
Inclusion Criteria:

* Initiation of antiretroviral therapy, consisting of 2 nucleoside/ nucleotide reverse transcriptase inhibitors at physician's disposition plus a third substance, i.e. either raltegravir (n=10 patients) or a standard third substance (efavirenz or boosted protease inhibitor)
* Men or women with a documented HIV-1 infection, treated at the study center
* age at least 18 years old
* physical examination and vital signs, according to the treating physician do not give any hint for a active AIDS-defining illness or other serious disease
* patients are naive to cART or in therapy interruption for at least 3 months
* last available HIV-1 RNA was >5,000 copies/mL within 3 months prior to cART initiation
* last available CD4-cell count showed at least 200 cells/µL within 3 months prior to cART initiation
* according to German-Austrian antiretroviral treatment recommendations, there is a given therapy indication

Exclusion Criteria:

* cART with other than the above mentioned drugs
* administration of concomitant drugs with relevant impact on antiretroviral's pharmacokinetics
* documented problems with patient visit- or medication-adherence
* any condition or disease requiring a medication that may interact relevantly with cART

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who begin cART in regular clinical routine with 2N(t)RTI plus either (n=10 patients) raltegravir or (n=10 patients) a boosted protease inhibitor/ alternatively an NNRTI as third substance will be offered to participate in this non-interventional study. Observation time is a period of 4 months after cART initiation.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2010-06; Primary Completion 2011-03 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Dynamical measurement of HIV-1 DNA-species extracted from whole blood-PBMCs | one year

SECONDARY OUTCOMES:
CD4 cell counts | one year
plasma-HIV-1 RNA | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Johann Wolfgang Goethe-University Hospital, Frankfurt am Main, Hesse, Germany

REFERENCES:
- [Result] Stephan C, Baldauf HM, Barry J, Giordano FA, Bartholomae CC, Haberl A, Bickel M, Schmidt M, Laufs S, Kaderali L, Keppler OT. Impact of raltegravir on HIV-1 RNA and DNA forms following initiation of antiretroviral therapy in treatment-naive patients. J Antimicrob Chemother. 2014 Oct;69(10):2809-18. doi: 10.1093/jac/dku213. Epub 2014 Jun 23. PMID 24962031
- Available data/document: Study Protocol: 01168167 — https://clinicaltrials.gov/ct2/show/NCT01168167